CLINICAL TRIAL: NCT03520465
Title: Utility of a Supraaponeurotic Mesh as Prophylaxis of the Midline Eventration After an Oncological Colorrectal Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PEACE
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Eventration
MeSH Terms: conditions — Gastroschisis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind, for the patient and the radiologist who analyses the results of the imaging tests.

ARMS (2):
- Supraaponeurotic mesh (Experimental): Patients with laparotomy closure by conventional approach of aponeurosis (continuous suture with monofilament of slow absorption), and posterior placement of supraaponeurotic mesh of polyvinylidene fluoride (PVDF) medium / low density and wide pore. The mesh has a longitudinal measurement that exceeds about 3 cm the upper and lower ends of the wound and width should not be less than 10 cm, therefore the mesh selected is DynaMesh®-CICAT longitudinal measure 10x35 cm.
  The mesh is fixed to the aponeurosis with a crown of loose stitches and points to the midline. A prolene 2/0 non-reabsorbable monofilament suture of cylindrical needle is used.
  A 10 Fr suction drainage is placed in the supraaponeurotic plane, with an exit to the exterior beyond the edges of the prosthesis. Drainage will be preserved for a minimum of 48 hours after surgery, and will be withdrawn when a debit of less than 50 ml is presented in 24 h.
  Interventions: Device: DynaMesh®-CICAT longitudinal measure 10x35 cm
- Monofilament (No Intervention): Patients with conventional closure of the middle laparotomy with approach of aponeurosis in a plane by continuous suture with monofilament of slow absorption. In this study, the suture used in all patients will be poly-4-hydroxybutyrate or Mono-max loop®.

INTERVENTIONS:
Device: DynaMesh®-CICAT longitudinal measure 10x35 cm
  Arms: Supraaponeurotic mesh

SUMMARY:
Randomized prospective experimental study, in which the effect of a prophylactic mesh is assessed in the eventration rate diagnosed by CT at one year after surgery in patients with CRC who underwent elective intervention for supra-infraumbilical midline laparotomy, considering as treatment the supra-aponeurotic mesh positioning (experimental group), and comparing it to the standard closing with a continuous suture using slow absorption monofilament.

DETAILED DESCRIPTION:
Randomized prospective experimental study, in which we evaluate patients with CRC who underwent elective intervention for supra-infraumbilical midline laparotomy in order to:

Main objective:

- To assess the effect of the prophylactic mesh in the eventration rate diagnosed by CT at one year after surgery in patients with CRC who underwent elective intervention for supra-infraumbilical midline laparotomy.

Secondary objectives:

* To compare the appearance of complications in the control group and in the experimental group.
* Compare costs derived from short and long-term mesh placement in both groups.

We consider as treatment the supra-aponeurotic mesh positioning (experimental group), and compare it to the standard closing with slow absorption monofilament.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery for colorectal cancer.
* Surgery by middle laparotomy.
* Informed consent signed by the patient.
* Age > 18 years.

Exclusion Criteria:

* Midline hernia or eventration.
* Presence of mesh in the abdominal wall because of a previous surgery.
* Palliative surgery.
* Synchronous metastases (Stage IV cancer according to TNM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2016-06-27 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Eventration rate | 1 year
  To assess the effect of the prophylactic mesh in the eventration rate diagnosed by CT at one year after surgery in patients with CRC who underwent elective intervention for supra-infraumbilical midline laparotomy.

SECONDARY OUTCOMES:
Complications rate | 1 year
  To compare the appearance of complications in the control group and in the experimental group.
Short and long term derived costs | 1 year
  To compare the costs derived from short and long-term mesh placement in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Frasson, Principal Investigator — Instituto de Investigación Sanitaria La Fe
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No